CLINICAL TRIAL: NCT00542438
Title: Feasibility and Validity of Home-Based Measures of Physical Activity and Body Composition
Brief Title: Home-Based Measures of Physical Activity and Body Composition
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-0278; NCI-2011-02917 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Cancer Prevention; Physical Activity; Body Composition; Environment; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Recall (Active Comparator): Hand-held computers will be used to record information for 7 days about physical activity. Assessments will be completed either 3 times a day or once a day.
  Interventions: Behavioral: Physical Activity Recall
- Environmental Assessment (Active Comparator): Environmental assessments on a palm pilot either 3 times a day or once a day. Hand-held computer programs will be used to collect information about the community. Some factors will be assessed only once (e.g., availability of facilities) while other information will be collected over the course of 7 days (e.g., perceptions of neighborhood safety).
  Interventions: Behavioral: Environmental Assessments

INTERVENTIONS:
Behavioral: Physical Activity Recall — Hand-held computers will be used to record information for 7 days about physical activity. Assessments will be completed either 3 times a day or once a day.
  Arms: Physical Activity Recall
Behavioral: Environmental Assessments — Hand-held computer programs will be used to collect information about the community. Some factors will be assessed only once (e.g., availability of facilities) while other information will be collected over the course of 7 days (e.g., perceptions of neighborhood safety).
  Arms: Environmental Assessment

SUMMARY:
The specific aim of this study is to collect preliminary data on the feasibility and validity of home-based data collection methods to measure four constructs:

* Physical Activity: Real-time assessment using Ecological Momentary Assessment (EMA) and pedometers
* Cardiorespiratory Fitness: Step test
* Anthropometry: Waist and hip circumference measurements
* Environmental Variables: Examples include density of neighborhood physical activity facilities (including gyms, parks, walking trails), crime, land use mix, and transportation variables, collected by participants using EMA.

DETAILED DESCRIPTION:
SCREENING PHONE CALL:

If you are interested in taking part in this study, the study staff will contact you by phone and you will answer questions about your physical ability to exercise. Based on the answers you give, the study doctor will decide if you are eligible to participate. The phone call will last about 10-15 minutes.

STUDY PROCEDURES:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to complete physical activity recall and environmental assessments on a palm pilot either 3 times a day or once a day. For the physical activity recall assessment, you will describe what types of physical activity you did that day. The environmental assessments will be to describe your current location or environment. It should take less than 5 minutes to complete each assessment.

Visit 1:

You will come to the M. D. Anderson Behavioral Research and Treatment Center for 2 visits. At the first visit, the following tests and procedures will be performed:

* Your height and weight will be measured.
* You will complete a questionnaire about your health, your neighborhood, and your physical activity. The questionnaire will take about 30 minutes to complete.
* You will walk on a treadmill while your heart rate, blood pressure, and respiration (breathing) are monitored. You will walk until you feel fatigued.

The research staff will then give you instructions for the tests you will do at home. This visit will last about 120 minutes.

At Home Activities:

During the next week, you will wear a pedometer and an actigraph. These are small devices that you wear on your waist during the day from the time you get up in the morning to when you go to bed at night. You will not wear the devices in water. These devices will record how active you are.

You will answer questions on a handheld computer 5-7 times each day. These questions will ask about your physical activity and about how your environment may encourage or discourage physical activity. It will take between 30 seconds and 3 minutes to answer the questions each time.

You will measure the distance around your waist and hips (circumference). You will do a fitness test that involves stepping up and down on a small stool for 3 minutes. You will take your heart rate after the stool-stepping exercise. The study staff will give you all the equipment and supplies needed for these tests at the first visit, and you will be asked to return the equipment at the second visit.

Visit 2:

Seven (7) days after the first visit, you will return to M. D. Anderson for the second visit. The following tests and procedures will be performed:

* You will perform the stool-stepping test.
* You will have your waist and hip circumference measured.
* You will be asked about your physical activity over the past week.

This visit will take about 60 minutes.

LENGTH OF STUDY:

You will be off-study once you complete Visit 2.

This is an investigational study. Up to 75 individuals will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. low-risk for cardiovascular disease, as defined by the American College of Sports Medicine (under 45 years of age for men and under 55 years of age for women, and less than two cardiovascular risk factors)
2. speaks English
3. able to give informed consent
4. no previous cancer diagnosis

Exclusion Criteria:

1. pregnant women
2. children under 18

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-10-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of home-based data collection methods: Percentage of Participants Completing Step Test | 3 Years
  Feasibility measured by the percentage of participants who have adequate cardiorespiratory fitness (i.e., V02 max greater than or equal to 31) to perform the step test. Researchers will consider the test feasible if greater than or equal to 75% of the participants have adequate fitness to perform the test.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org